CLINICAL TRIAL: NCT00106548
Title: A Randomized, Double-blind Study of Safety and Reduction in Signs and Symptoms During Treatment With Tocilizumab Versus Placebo, in Combination With Methotrexate, in Patients With Moderate to Severe Rheumatoid Arthritis
Brief Title: A Study to Assess the Effect of Tocilizumab + Methotrexate on Signs and Symptoms in Patients With Moderate to Severe Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Clinical Trials, Study Director, Hoffmann-La Roche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WA17822
Record Dates: First submitted 2005-03-25; First posted 2005-03-28 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]; Drug: Methotrexate
- 2 (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]; Drug: Methotrexate
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Methotrexate

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — 4mg/kg iv / month
  Arms: 1
Drug: tocilizumab [RoActemra/Actemra] — 8mg/kg iv / month
  Arms: 2
Drug: Placebo — iv / month
  Arms: 3
Drug: Methotrexate — 10-25mg/week

SUMMARY:
This 3 arm study will compare the safety and efficacy, with regard to reduction of signs and symptoms, of tocilizumab versus placebo, both in combination with methotrexate (MTX). in patients with moderate to severe active rheumatoid arthritis (RA) who currently have an inadequate response to MTX. Patients wil be randomized to receive tocilizumab 4mg/kg iv, tocilizumab 8mg/mg iv, or placebo iv, every 4 weeks; all patients will also receive methotrexate 10-25mg weekly. The anticipated time on study treatment is 3-12 months, and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients at least 18 years of age with moderate to severe active RA for at least 6 months;
* inadequate response to a stable dose of MTX;
* patients of reproductive potential must be using reliable methods of contraception.

Exclusion Criteria:

* major surgery (including joint surgery) within 8 weeks before entering study, or planned surgery within 6 months after entering study;
* prior treatment failure with an anti-tumor necrosis factor agent;
* women who are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 623 (Actual)
Dates: Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with ACR 20 response | Week 24

SECONDARY OUTCOMES:
Percentage of patients ACR 50/70 responses; change from baseline in ACR core set components. | Week 24
AEs, laboratory parameters, vital signs | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (59):
- Buenos Aires, Argentina
- Australia (4):
  - Adelaide
  - Douglas
  - Maroochydore
  - Shenton Park
- Vienna, Austria
- Brazil (2):
  - Porto Alegre
  - São Paulo
- Bulgaria (2):
  - Sofia
  - Varna
- Canada (11):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - St. John's, Newfoundland and Labrador
  - Burlington, Ontario
  - Newmarket, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Sainte-Foy, Quebec
- Hong Kong, China
- France (5):
  - Besançon
  - Créteil
  - Le Mans
  - Montpellier
  - Paris
- Germany (8):
  - Bad Bramstedt
  - Bad Nauheim
  - Baden-Baden
  - Berlin
  - Cologne
  - Erlangen
  - Heidelberg
  - Tübingen
- Hungary (3):
  - Budapest
  - Debrecen
  - Pécs
- Israel (5):
  - Beersheba
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Tel Aviv
- Italy (5):
  - Ferrara
  - Gazzi
  - Palermo
  - Siena
  - Udine
- Mexico (4):
  - Chihuahua City
  - Guadalajara
  - Mexico City
  - San Luis Potosí City
- Singapore, Singapore
- Piešťany, Slovakia
- Switzerland (3):
  - Bern
  - Lausanne
  - Sankt Gallen
- Thailand (2):
  - Bangkok
  - Chiang Mai

REFERENCES:
- [Derived] Keystone EC, Anisfeld A, Ogale S, Devenport JN, Curtis JR. Continued benefit of tocilizumab plus disease-modifying antirheumatic drug therapy in patients with rheumatoid arthritis and inadequate clinical responses by week 8 of treatment. J Rheumatol. 2014 Feb;41(2):216-26. doi: 10.3899/jrheum.130489. Epub 2014 Jan 15. PMID 24429164
- [Derived] Wang J, Bansal AT, Martin M, Germer S, Benayed R, Essioux L, Lee JS, Begovich A, Hemmings A, Kenwright A, Taylor KE, Upmanyu R, Cutler P, Harari O, Marchini J, Criswell LA, Platt A. Genome-wide association analysis implicates the involvement of eight loci with response to tocilizumab for the treatment of rheumatoid arthritis. Pharmacogenomics J. 2013 Jun;13(3):235-41. doi: 10.1038/tpj.2012.8. Epub 2012 Apr 10. PMID 22491018
- [Derived] Garnero P, Thompson E, Woodworth T, Smolen JS. Rapid and sustained improvement in bone and cartilage turnover markers with the anti-interleukin-6 receptor inhibitor tocilizumab plus methotrexate in rheumatoid arthritis patients with an inadequate response to methotrexate: results from a substudy of the multicenter double-blind, placebo-controlled trial of tocilizumab in inadequate responders to methotrexate alone. Arthritis Rheum. 2010 Jan;62(1):33-43. doi: 10.1002/art.25053. PMID 20039425
- [Derived] Smolen JS, Beaulieu A, Rubbert-Roth A, Ramos-Remus C, Rovensky J, Alecock E, Woodworth T, Alten R; OPTION Investigators. Effect of interleukin-6 receptor inhibition with tocilizumab in patients with rheumatoid arthritis (OPTION study): a double-blind, placebo-controlled, randomised trial. Lancet. 2008 Mar 22;371(9617):987-97. doi: 10.1016/S0140-6736(08)60453-5. PMID 18358926